CLINICAL TRIAL: NCT05360615
Title: The Effects of Empagliflozin on Renal Outcomes in Post Severe Acute Kidney Injury Survivors
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Chulalongkorn University (Other)
Responsible Party: Principal Investigator, Nattachai Srisawat ,M.D., Assistant Professor.Nattachai Srisawat, Chulalongkorn University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB.211/65
Record Dates: First submitted 2022-04-30; First posted 2022-05-04 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: Empagliflozin in Post AKI Stage 2-3
Keywords: Empagliflozin; AKI
MeSH Terms: interventions — empagliflozin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Empagliflozin (Experimental)
  Interventions: Drug: Empagliflozin 10 MG
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Empagliflozin 10 MG — SGLT2 inhibitors
  Arms: Empagliflozin
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
Effects of Empagliflozin compared with placebo in post severe acute kidney injury survivors, evaluated by MAKE365.

ELIGIBILITY:
Inclusion Criteria:

* post AKI stage 2-3
* CrCl > 20

Exclusion Criteria:

* pregnancy
* post kidney transplant
* previous use of SGLT2 Inhibitors
* history of ketoacidosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 147 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
MAKE365 | 1 year
  Major adverse kidney events (number of participants with death, renal replacement therapy, New CKD, CKD progression)

CONTACTS AND LOCATIONS:
Overall Officials: Nattachai Srisawat, Principal Investigator — Chulalongkorn University
Locations (1):
- Central Chest Institute of Thailand, Nonthaburi, Mueang Nonthaburi District, Thailand

IPD SHARING:
Plan to Share IPD: Undecided